CLINICAL TRIAL: NCT06134687
Title: Prospective Single Centre, Post Market, Randomized Controlled Trial to Demonstrate Feasibility, Safety and Efficacy, of a Novel Rigidizing Overtube in Colonic Endoscopic Submucosal Dissection
Brief Title: Novel Rigidizing Overtube in Colonic Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Neptune Medical, Inc. (Unknown)
Responsible Party: Principal Investigator, Mohamed Othman, MD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-53924
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment arm (Experimental): Will have endoscopic submucosal dissection performed with the use of the Pathfinder Endoscope Overtube.
  Interventions: Procedure: Endoscopic Submucosal Dissection; Device: Novel Rigidizing Overtube
- Control arm (Active Comparator): Will have endoscopic submucosal dissection performed through conventional means (i.e. without the Pathfinder Endoscope Overtube).
  Interventions: Procedure: Endoscopic Submucosal Dissection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Removal of study eligible lesions per endoscopic submucosal dissection
  Other Names: ESD; Endoscopic resection
Device: Novel Rigidizing Overtube — Utilization of the Novel Rigidizing Overtube (Pathfinder) to aid in performing colonic endoscopic submucosal dissection
  Arms: Treatment arm

SUMMARY:
The goal of this prospective, single centre, 1:1, Post Market, randomized controlled, Investigator Initiated trial, is to compare the feasibility, safety efficacy, and clinical outcomes of colonic endoscopic submucosal dissection (ESD) utilizing a novel rigidizing overtube called Pathfinder® Endoscope Overtube (Neptune Medical, Burlingame California, USA) device in comparison to conventional ESD.

The research team hypothesize that with utilizing a novel rigidizing overtube the procedure time including dissection speed and closure time will be faster due to higher scope stability and greater control over the scope tip. Subsequently, the investigators anticipate lower immediate or delayed adverse events.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is preferred resection method for advanced colonic polyp due to its higher rates of en bloc and R0 resection which lead to higher curative resection rate.1 In comparison to gastric ESD, colonic ESD is more challenging due to colonic unique anatomy and configuration. Tumor of size ≥ 50 mm, spreading across ≥ two folds, flexure locations have been described as strong predictors for difficulties during colonic ESD.2 Redundant colon and looping during colonoscopy may preclude successful advancement of the colonoscope and maintaining stable position for complex polyp removal.

Historically, various methods have been applied to facilitate colonoscopy and scope advancement in challenging positions and redundant colonic loops such as application of external pressure, exchange to pediatric colonoscope, torque-based reduction maneuvers, and patient repositioning. However, despite these, scope tip stabilization could potentially remain as a challenging and limiting factor for procedure progress and could lead to a longer procedure time, sedation time and perhaps lower procedure success rate. In comparison overtube-assisted colonoscopy allows for straightening of the colon to decrease angulation and loop formation.3 Several variations of overtubes have been put to use in the last few decades with comparable results such as single-balloon and double-balloon enteroscope, spiral overtube-assisted colonoscopy and double-balloon platform (DiLumenTM). DiLumen system consists of a plastic sheet fitting layer with two balloon few inches from each other in the tip of the device facilitating the scope tip stability. Most recently the efficacy of DiLumen platform were evaluated in a multicenter study including 162 patients who underwent endoscopic resection of advanced polyps.4 In this study technical success was achieved in 92% of patients without any device related adverse event. 4 In this study using an overtube resulted in faster and more efficient dissection.4 In a retrospective study of 88 polyps located within the proximal colon, ESD with assistance of traditional single balloon overtube resulted in significantly less perforation rate in polyps ≥ 40mm in the proximal colon, despite overall similar en bloc and R0 resection rates comparison to conventional ESD.5 Most recently, a novel dynamic rigidizing overtube (Pathfinder, Neptune Medical, Burlingame, Calif, USA) has been introduced to face the challenges encountered during difficult colonoscopies and to ensure scope stabilization during endoscopic mucosal resection (EMR) and ESD. The overtube material is soft and pliable on flexible state, however when the vacuum is applied the entire tube becomes 15 times stiffer.6 This unique feature of the device provides scope flexibility during colonoscope introduction and entire device stability when rigidizing system is applied.

Our team collected preliminary prospective data of 58 polyps removed by EMR (24.1%) and ESD (75.9% ) with the assistance off rigidizing overtube. Technical success (ability to complete the entire resection using the device) and clinical success (ability of endoscopic removal of polyps without changing the initial resection intent) was achieved 100% and 90% of the time, respectively. On endoscopist feedback, the rigidizing overtube was though to assist in resection in 98.3% of polyps, although the polyp was located in a somewhat/very difficult location 81% of the time. For polyps in difficult locations, the rigidizing overtube was able to maintain scope position without falling back even once, 55% of the time. This result was presented at the most recent Digestive Disease Week conference in Chicago 2023 (p1932).

As this device has been put to use recently in the United States, published literature to demonstrate its safety and efficacy in colonic ESD is lacking. The main aim of this study is to compare the feasibility, safety efficacy, and clinical outcomes of colonic endoscopic submucosal dissection (ESD) utilizing a novel rigidizing overtube called Pathfinder® Endoscope Overtube (Neptune Medical, Burlingame CA, USA) device in comparison to conventional ESD.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 22 years old.
* Patients can provide written informed consent.
* Patient is referred for ESD procedure of colonic neoplastic lesions and with one of the following criteria:

A - Lesions with prior resection or with scar at any size proximal to the sigmoid colon.

B - Granular lateral spreading tumors (GLST) more than 30mm. C - Non granular lateral spreading tumors (NGLST) more than 20 mm. D - Any suspected submucosal invasion such as Paris classification II a +II or lesions with positive non lifting sign.

Exclusion Criteria:

* Patient refused and/or unable to provide written informed consent.
* Patient is a pregnant or nursing woman.
* Lesions with morphology: pedunculated type (Paris Ip, Ips).
* Lesions located within the sigmoid colon or rectum.
* Lesions involving appendiceal orifice or ileocecal valve

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Total Procedure Time | Day 1 (procedure day)
  Total Procedure Time to perform ESD from scope in to scope out

SECONDARY OUTCOMES:
Navigation Time | Day 1 (procedure day)
  Total time needed to reach the lesion
Technical Success | Day 1 (procedure day)
  The ability to complete the entire resection using the device without the need to change to a different tool. This will be marked as either 'yes' or 'no' on the collection report form following the procedure by the research team.
Clinical Success | Day 1 (procedure day)
  The ability of endoscopic removal of polyps without changing the initial resection intent. This will be marked as either 'yes' or 'no' on the collection report form following the procedure by the research team.
En-bloc, R0, and curative resection rates | Day 1 (procedure day)
  As collected and measured for each group
Dissection speed during colonic ESD as calculated by | Day 1 (procedure day)
  cm^2/hr
Closure time | Day 1 (procedure day)
  Time needed to close area following endoscopic resection
Sedation time | Day 1 (procedure day)
  Total time patient spent under anesthesia
User-feedback post-procedure | Day 1 (procedure day)
  Subjective assessment of the degree of difficulty reaching the lesion based on a brief questionnaire given to the endoscopist following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Lukes Medical Center (BSLMC), Houston, Texas